CLINICAL TRIAL: NCT07028697
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel, Phase III Study to Evaluate the Efficacy and Safety of ACT-541468 (Daridorexant) in Adult and Elderly Subjects With Insomnia Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Daridorexant in Participants With Insomnia Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nxera Pharma Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPK-DAR-301
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daridorexant (Experimental)
  Interventions: Drug: Daridorexant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant — Daridorexant will be taken orally, once daily in the evening as indicated by investigator.
  Arms: Daridorexant
Drug: Placebo — Placebo will be taken orally, once daily in the evening as indicated by investigator.
  Arms: Placebo

SUMMARY:
The purpose of this phase 3 study is to evaluate the efficacy and safety of Daridorexant compared to in participants with insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure;
* Male or female aged ≥ 19 years;
* Insomnia disorder according to DSM-5 criteria;
* The predominant complaint is dissatisfaction with sleep quantity or quality, associated with one (or more) of the following symptoms:
* Difficulty initiating sleep.
* Difficulty maintaining sleep (characterized by frequent awakenings or problems returning to sleep after awakenings).
* Early-morning awakening with inability to return to sleep.
* Insomnia Severity Index score ≥ 15;
* Insufficient sleep quantity as collected subjectively in the sleep diary A. ≥ 30 min to fall asleep, and B. Wake time during sleep ≥ 30 min, and C. Subjective Total Sleep Time (sTST) ≤ 6.5 h

Exclusion Criteria:

* Body mass index (BMI) ≥ 40.0 kg/m2
* Documented medical history and/or comorbidity of sleep-related breathing disorder
* History of and/or concurrent sleep apnea or suspected sleep apnea
* Korean-Mini Mental State Examination-2 (K-MMSE-2) score < 25 in subjects ≥ 50 years;
* For female subjects: pregnant, lactating or childbearing potential who do not consent to true abstinence or use an effective method of contraception for required period
* Initiation of the cognitive behavior therapy (CBT) for treatment of insomnia disorder within 4 weeks prior to the Screening visit (Visit 1) or planned CBT during the study
* A history of moderate to severe hepatic impairment (eg, Child-Pugh Class B or C)
* Positive urine drug test or presence of alcohol in exhaled breath as detected by breathalyzer test.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Subjective total sleep time(sTST) | Week 4
  Change from baseline to week 4 in subjective total sleep time (sTST) measured by eDairy

SECONDARY OUTCOMES:
Subjective latency to sleep onset (sLSO) | Week 4
  Change from baseline to week 4 in subjective latency to sleep onset (sLSO) measured by eDairy
Subjective wake after sleep onset (WASO) | Week 4
  Change from baseline to week 4 in subjective wake after sleep onset (WASO) measured by eDairy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Nxera Pharma Korea Co., Ltd., Study Director — Nxera Pharma Korea Co., Ltd.
Locations (17):
- South Korea (17):
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Catholic Kwandong University International St. Mary'S Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyung Hee University Hospital At Gangdong, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Medical Center, Seoul
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju